CLINICAL TRIAL: NCT00002756
Title: Induction Intensification in Infant ALL: A Children's Oncology Group Study
Brief Title: Induction Intensification in Treating Infants With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P9407; COG-P9407 (Other: Children's Oncology Group); POG-9407 (Other: Pediatric Oncology Group); CDR0000064693 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia; acute undifferentiated leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Biphenotypic, Acute | interventions — Filgrastim; Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Etoposide; Leucovorin; Mercaptopurine; Methotrexate; Prednisone; Hydrocortisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemo (Reduced Induction) No BMT (Open February 2004) (Experimental)
  Interventions: Biological: filgrastim; Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: etoposide; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: filgrastim
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: etoposide
Drug: leucovorin calcium
Drug: mercaptopurine
Drug: methotrexate
Drug: prednisone
Drug: therapeutic hydrocortisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one chemotherapy drug and giving them as induction intensification may kill more cancer cells.

PURPOSE: This phase II trial is studying how well induction intensification works in treating infants with newly diagnosed acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the feasibility of intensification with two courses of high-dose methotrexate followed by one course of cyclophosphamide/etoposide during induction and later as consolidation in infants with newly diagnosed acute lymphoblastic leukemia.
* Determine event-free survival after shortened, intensive therapy in these patients.
* Compare event-free survival rates of infants receiving this regimen whose leukemic blasts have or do not have translocations involving the 11q23 gene MLL.

Secondary

* Correlate the presence of minimal residual disease at completion of induction, beginning of continuation, and at completion of therapy with patient outcome.
* Investigate the clinical prognostic features that may be associated with outcome in infants, such as bone marrow blast content at day 8, white blood cell count, and age.
* Correlate biologic characteristics of the leukemia cells at diagnosis (protocol POG-9900) with outcome in patients treated with this regimen.
* Characterize patterns of gene expression associated with host and disease characteristics and treatment response in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center and presence of CNS disease (yes vs no).

Patients receive induction chemotherapy comprising vincristine IV on days 1, 8, and 15; oral prednisone three times a day on days 1-21; daunorubicin IV over 30 minutes on days 1-2; cyclophosphamide IV over 30 minutes every 12 hours on days 3-4; and asparaginase intramuscularly (IM) on days 4, 6, 8, 10, 12, 15, 17, and 19. Patients also receive triple intrathecal therapy comprising methotrexate, hydrocortisone, and cytarabine on days 1, 8, and 15 and filgrastim (G-CSF) subcutaneously (SC) or IV beginning on day 5 and continuing until day 20, regardless of blood counts.

Patients receive induction intensification chemotherapy comprising high-dose methotrexate IV over 24 hours; triple intrathecal therapy as per induction therapy on days 22 and 29; and leucovorin calcium IV every 6 hours for 2 doses beginning 42 hours after start of high-dose methotrexate and then orally every 6 hours for 3 doses. Patients also receive etoposide IV over 2 hours and cyclophosphamide IV over 30 minutes on days 36-40. Patients receive G-CSF SC or IV beginning on day 41 and continuing until blood counts recover.

Patients achieving morphologic remission and recovery of blood counts while off G-CSF for 48 hours receive reinduction chemotherapy comprising the same regimen as in induction therapy with the exception of asparaginase IM beginning on day 1 (week 8) and continuing every Monday, Wednesday, and Friday for a total of 8 doses and triple intrathecal therapy on days 1 and 15 only (weeks 8 and 10). Patients receive G-CSF SC or IV beginning on day 5 and continuing until blood counts recover.

After blood count recovery, patients receive consolidation chemotherapy comprising triple intrathecal therapy as per induction therapy on day 1 (week 11); high-dose methotrexate IV over 24 hours on weeks 8 and 12; and leucovorin calcium IV every 6 hours for 2 doses beginning 42 hours after start of high-dose methotrexate and then orally every 6 hours for 3 doses. Patients also receive etoposide IV over 2 hours followed by cyclophosphamide IV over 30 minutes on days 15-19 (week 13). Patients receive G-CSF SC or IV beginning on day 20 and continuing until blood counts recover. On days 29-31 (week 15), patients receive high-dose cytarabine IV over 3 hours every 12 hours for 4 doses and asparaginase IM 6 hours after completion of high-dose cytarabine. Patients receive G-CSF beginning 24 hours after completion of asparaginase and continuing until blood counts recover.

Patients achieving morphologic remission and blood count recovery while off G-CSF for 48 hours receive continuation therapy comprising vincristine IV on day 1; oral prednisone three times a day on days 1-5; and triple intrathecal therapy on day 1 (weeks 18 and 22). Patients also receive methotrexate IM once a week and oral mercaptopurine daily on weeks 19-21, 23, and 24. On week 25, patients receive etoposide IV over 2 hours daily followed by cyclophosphamide IV over 30 minutes daily on days 1-5 and G-CSF SC or IV beginning on day 6 and continuing until blood counts recover. Patients receive an additional course of continuation therapy on weeks 28-35. On weeks 38-48, patients receive another identical course of continuation therapy with the exclusion of the etoposide and cyclophosphamide combination regimen.

Patients are followed monthly for 1 year, every 2 months for 1 year, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 58-104 patients will be accrued for this study within 2.1 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute lymphoblastic leukemia (ALL) or acute undifferentiated leukemia

  * No infants less than 36 weeks' gestation
  * CNS or testicular disease permitted
* No B-cell ALL or acute myeloid leukemia
* Previously untreated except for the following:

  * Steroid treatment within 48 hours of diagnosis allowed with physical examination and differential CBC immediately prior to beginning steroids
* Concurrent registration on protocol POG-9900 (ALL classification study) required
* Patients registered on POG-9407 are eligible for the pharmacokinetic part of the study

PATIENT CHARACTERISTICS:

Age:

* Under 1 at diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No uncontrolled infection
* Adequate major organ function

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* See Disease Characteristics
* No concurrent chronic steroid treatment

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No other concurrent anticancer therapy

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 221 (Actual)
Dates: Start 1996-06; Primary Completion 2007-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of intensification
Event-free survival
Comparison of event-free survival rates in infants with and without leukemic blasts translocations

SECONDARY OUTCOMES:
Correlation of minimal residual disease at completion of induction, beginning of continuation, and at completion of therapy with patient outcome
Clinical prognostic features associated with outcome
Correlation of biologic characteristics of leukemia cells at diagnosis with outcome
Patterns of gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Zoann E. Dreyer, MD, Study Chair — Texas Children's Cancer Center
Locations (140):
- United States (128):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center - Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Children's Hospital, Santa Barbara, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center - Fairview, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - INOVA Fairfax Hospital, Fairfax, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Cancer Center of Western Virginia, Roanoke, Virginia
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Background] Dreyer ZE, Dinndorf PA, Camitta B, Sather H, La MK, Devidas M, Hilden JM, Heerema NA, Sanders JE, McGlennen R, Willman CL, Carroll AJ, Behm F, Smith FO, Woods WG, Godder K, Reaman GH. Analysis of the role of hematopoietic stem-cell transplantation in infants with acute lymphoblastic leukemia in first remission and MLL gene rearrangements: a report from the Children's Oncology Group. J Clin Oncol. 2011 Jan 10;29(2):214-22. doi: 10.1200/JCO.2009.26.8938. Epub 2010 Dec 6. PMID 21135279
- [Background] Fernandez CV, Kodish E, Taweel S, Shurin S, Weijer C; Children's Oncology Group. Disclosure of the right of research participants to receive research results: an analysis of consent forms in the Children's Oncology Group. Cancer. 2003 Jun 1;97(11):2904-9. doi: 10.1002/cncr.11391. PMID 12767106
- [Result] Kang H, Wilson CS, Harvey RC, Chen IM, Murphy MH, Atlas SR, Bedrick EJ, Devidas M, Carroll AJ, Robinson BW, Stam RW, Valsecchi MG, Pieters R, Heerema NA, Hilden JM, Felix CA, Reaman GH, Camitta B, Winick N, Carroll WL, Dreyer ZE, Hunger SP, Willman CL. Gene expression profiles predictive of outcome and age in infant acute lymphoblastic leukemia: a Children's Oncology Group study. Blood. 2012 Feb 23;119(8):1872-81. doi: 10.1182/blood-2011-10-382861. Epub 2011 Dec 30. PMID 22210879
- [Result] Salzer WL, Jones TL, Devidas M, Hilden JM, Winick N, Hunger S, Carroll WL, Camitta B, Dreyer ZE. Modifications to induction therapy decrease risk of early death in infants with acute lymphoblastic leukemia treated on Children's Oncology Group P9407. Pediatr Blood Cancer. 2012 Nov;59(5):834-9. doi: 10.1002/pbc.24132. Epub 2012 Apr 5. PMID 22488662
- [Result] Robinson BW, Devidas M, Carroll AJ, et al.: Specific MLL partner genes in infant acute lymphoblastic leukemia (ALL) associated with outcome are linked to age and white blood cell count (WBC) at diagnosis: A report on the Children's Oncology Group (COG) P9407 trial. [Abstract] Blood 114 (22): A-907, 2009.
- [Result] Thompson PA, Murry DJ, Rosner GL, Lunagomez S, Blaney SM, Berg SL, Camitta BM, Dreyer ZE, Bomgaars LR. Methotrexate pharmacokinetics in infants with acute lymphoblastic leukemia. Cancer Chemother Pharmacol. 2007 May;59(6):847-53. doi: 10.1007/s00280-006-0388-1. Epub 2006 Nov 29. PMID 17136402